CLINICAL TRIAL: NCT02023762
Title: Safety and Feasibility of Deep Sedation Instead of General Anaesthesia in Percutaneous Mitral Valve Repair Using the MitraClip® System
Brief Title: Deep Sedation Instead of General Anaesthesia in Percutaneous Mitral Valve Repair Using the MitraClip® System
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Director Division of Cardiology, Pulmonary Disease and Vascular Medicine, Heinrich-Heine University, Duesseldorf
Other Study IDs: MitraClip under sedation
Record Dates: First submitted 2013-12-12; First posted 2013-12-30 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Mitral Regurgitation; Local Anaesthesia; Percutaneous Repair
Keywords: mitral regurgitation; local anaesthesia; percutaneous repair
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Percutaneous mitral valve repair (PMVR) with the MitraClip® system has emerged as a therapeutic alternative to surgical valve repair in patients who are at high risk and unsuitable for surgery. The PMVR procedure is typically performed under general anaesthesia, but the MitraClip® is also feasible in deep sedation.

The aim of this study is to investigate the safety of deep sedation in patients undergoing the PMVR procedure and to evaluate how deep sedation in comparison to general anaesthesia influences procedural time and in-hospital stay.

DETAILED DESCRIPTION:
Percutaneous mitral valve repair (PMVR) with the MitraClip® system has emerged as a therapeutic alternative to surgical valve repair in patients who are at high risk and unsuitable for surgery.

The PMVR procedure, however, is typically performed under general anaesthesia. It has recently been shown in a first approach that performing the MitraClip® in deep sedation is feasible; however safety parameters and a direct comparison to general anaesthesia are still missing The aim of this study is to investigate the safety of deep sedation in patients undergoing the PMVR procedure and to evaluate how deep sedation in comparison to general anaesthesia influences procedural time and in-hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* severe mitral regurgitation
* PMVR using the MitraClip® system

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe mitral regurgitation characterized by trans-thoracic and trans-esophageal echocardiography undergoing PMVR using the MitraClip® system
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse Events | patients will be followed for the duration of procedure until discharge, an expected average of 10 days
  Evaluation of feasibility and safety of deep sedation instead of general anaesthesia

SECONDARY OUTCOMES:
preparation and procedure time | procedure
Overall time to discharge | Participants will be followed for the duration of hospital stay, an expected average of 10 days
Changes in 6-Minute Walk Test | Baseline to 1 month after intervention
Changes in NYHA class | Baseline to 1 month after intervention
Changes in N-terminal prohormone of brain natriuretic peptide (NT-proBNP) | Baseline to 1 month after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Tienush Rassaf, MD, Principal Investigator — Division of Cardiology, Pulmonary Disease and Vascular Medicine, University Hospital Dusseldorf; Malte Kelm, MD, Study Chair — Division of Cardiology, Pulmonary Disease and Vascular Medicine, University Hospital Dusseldorf

REFERENCES:
- [Derived] Rassaf T, Balzer J, Zeus T, Rammos C, Shayganfar S, Hall SV, Wagstaff R, Kelm M. Safety and efficacy of deep sedation as compared to general anaesthesia in percutaneous mitral valve repair using the MitraClip system. Catheter Cardiovasc Interv. 2014 Oct 1;84(4):E38-42. doi: 10.1002/ccd.25570. Epub 2014 Jul 4. PMID 24909413
- See also: Related Info — http://www.uniklinik-duesseldorf.de/kardiologie